CLINICAL TRIAL: NCT06434688
Title: Examining Mental Fatigue, Body Awareness, and Mindfulness in People With Chronic Neck Pain
Brief Title: Body Awareness and Mental Fatigue in Neck Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Selenay Aydogdu, principal Investigator, Hacettepe University
Other Study IDs: 10557444
Record Dates: First submitted 2024-05-09; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-02

CONDITIONS: Neck Pain; Mental Fatigue; Mindfulness; Awareness
Keywords: mental fatigue; Mindfulness; Interoception; Proprioception
MeSH Terms: conditions — Neck Pain; Mental Fatigue | interventions — Quality of Life; Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals experiencing neck pain: Study Group Inclusion Criteria:
  * Having chronic neck pain for at least 3 months.
  * Being between 18 and 65 years of age.
  * Scoring 5 and above on the Neck Disability Questionnaire.
  * Scoring 24 and above on the Mini Mental Status Examination.
  * Being able to read and write.
  * Being willing to participate in the study.
  Study Group Exclusion Criteria:
  * Participation in any physical therapy program in the last 3 months.
  * Having the following problems:
  * Radiculopathy, myleopathy (motor and sensory loss) and other neurologic diseases.
  * Inflammatory diseases
  * History of malignancy.
  * Congenital spinal cord anomaly and congenital spinal deformities
  * Spinal pathologies, traumatic medulla spinalis injury and other medulla spinalis pathologies.
  * Vestibular disorders.
  * Diagnosed psychiatric disorders such as bipolar disorder and panic attacks.
  * Vision problems that do not improve despite vision aids.
  * Pregnancy
  Interventions: Other: Mental Fatigue:; Other: Body Awareness:; Other: Neck Disability Level; Other: Quality Of Life; Other: Pain Assessment:; Other: Physical Condition:; Other: Anxiety and Depression:
- Healthy individuals without neck pain: Control Group Inclusion Criteria:
  * Age between 18 and 65 years.
  * Scoring 24 and above on the Mini Mental State Examination.
  * To be able to read and write.
  * Volunteering to participate in the study.
  Control Group Exclusion Criteria:
  * Having chronic pain in the spine, especially in the neck.
  * Exclusion criteria for the study group
  Interventions: Other: Mental Fatigue:; Other: Body Awareness:; Other: Quality Of Life; Other: Physical Condition:; Other: Anxiety and Depression:

INTERVENTIONS:
Other: Mental Fatigue: — The Mental Fatigue Scale (MFS) will be used to assess mental fatigue.
Other: Body Awareness: — Individuals' general body awareness will be assessed with the Body Awareness Questionnaire (BAQ).
  Neck awareness of individuals will be assessed with the Fremantle Neck Awareness Questionnaire (FreBFA).
  Short Form of the Five Facet Mindfulness Questionnaire (FFMQ - Short Form) will be used to assess people's mindfulness.
  - In-body awareness:
  For the sense of interoception, the Multidimensional Assessment of Interoceptive Awareness Scale, which assesses interoceptive body awareness, will be used.
  To evaluate proprioception, a Cervical Range of Motion (CROM) device is used.
  The bucket test will be used to assess subjective visual verticality, which is one of the sub-dimensions of verticality perception.
  Two scales will be used to assess people's awareness of weight transfer symmetry.
  - Out of Body Awareness:
  "Right-Left Confusion Hand Test" will be used to evaluate the mental rotation skill within the scope of the sense of extroception.
Other: Neck Disability Level — Neck disability index will be used to assess this parameter.
  Groups: Individuals experiencing neck pain
Other: Quality Of Life — SF-12 will be used to assess quality of life.
Other: Pain Assessment: — Pain intensity will be assessed by Visual Analog Scale (VAS). In addition, pain duration and pain frequency will be questioned. The Pain Self-Efficacy Questionnaire will be used to assess the confidence of people with chronic pain to perform certain tasks and behaviors despite their pain.
  Groups: Individuals experiencing neck pain
Other: Physical Condition: — Normal range of motion of the cervical region will be evaluated with the "Cervical Range of Motion" device.
  New York Posture Rating Scale will be used to evaluate posture.
  Symmetry of weight transfer to both lower extremities of the individuals in standing upright position will be evaluated.
Other: Anxiety and Depression: — Beck Depression and Beck Anxiety scales will be used to assess depression and anxiety.

SUMMARY:
The primary aim of the study was to examine the difference between mental fatigue, in-body, out-of-body and mindfulness parameters in people with chronic neck pain compared to a healthy control group, and to analyze the relationships between mental fatigue and neck disability level and awareness levels, and between awareness levels and neck disability level and quality of life.

The secondary aim was to examine the relationships between pain intensity, frequency, duration, pain self-efficacy, physical condition, anxiety and depression, mental fatigue and awareness levels in people with chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is a prevalent musculoskeletal issue that can cause significant disability. Individuals with neck pain may experience changes in muscle structure and behavior, as well as sensory-perceptual-motor issues such as decreased proprioception and related neuromuscular changes. Additionally, neck pain can lead to psychological problems such as anxiety and depression.Although some awareness parameters have been evaluated in studies on neck pain in the literature and it has been shown that chronic pain is associated with impaired body awareness and that this impairment contributes to and/or maintains chronic pain, no study has been found to examine all awareness parameters in detail. Another cause that compromises the accuracy of information contributing to body awareness is mental fatigue. Mental fatigue can negatively affect a person's level of perception. In one study, it was stated that mental fatigue was a determinant of neck disability, but studies on this subject were found to be very insufficient. Therefore, the aim of this study was to examine the sub-parameters of awareness and mental fatigue in people with chronic neck pain, to compare them with healthy people and to examine the relationship between the parameters evaluated.

ELIGIBILITY:
Study Group Inclusion Criteria:

* Having chronic neck pain for at least 3 months.
* Being between 18 and 65 years of age.
* Scoring 5 and above on the Neck Disability Questionnaire.
* Scoring 24 and above on the Mini Mental State Examination.
* To be able to read and write.
* Being volunteer to participate in the study.

Study Group Exclusion Criteria:

* Participation in any physical therapy program in the last 3 months.
* Having the following problems:
* Radiculopathy, myleopathy (motor and sensory loss) and other neurological diseases.
* Inflammatory diseases (rheumatoid arthritis, etc.).
* History of malignancy.
* Congenital spinal cord anomaly and congenital spinal deformities.
* Spinal pathologies, traumatic medulla spinalis injury and other medulla spinalis pathologies.
* Vestibular disorders.
* Diagnosed psychiatric illnesses such as bipolar disorder, psychotic illnesses and panic attacks.
* Vision problems that do not fully recover despite vision aids (glasses, etc.).
* Pregnancy status

Control Group Inclusion Criteria:

* Age between 18 and 65 years.
* Scoring 24 and above on the Mini Mental State Examination.
* To be able to read and write.
* Volunteering to participate in the study.

Control Group Exclusion Criteria:

* Having chronic pain in the spine, especially in the neck.
* Exclusion criteria for the study group

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with neck pain and healthy individuals without neck pain
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2024-05-27 (Estimated); Primary Completion 2024-07-29 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Mental Fatigue | 2024 may- 2024 July
  The Mental Fatigue Scale (MFS) will be used to assess mental fatigue. It includes questions about general fatigue, lack of initiative, mental fatigue, concentration difficulties, memory problems, slowness of thinking, sensitivity to stress, increased tendency to be emotional, irritability, sensitivity to light and noise, decreased or increased sleep. It has a 7-point Likert-type scale and is scored from 0 to 3. A rating of 0 indicates normal functioning, 1 indicates mild problem, 2 indicates significant problem and 3 indicates maximum problem. According to the total score, 0-10= no mental fatigue problem, 10.5-14.5= mild mental fatigue, 15-20= quite serious mental fatigue, ≥ 20.5= serious mental fatigue.
General Body Awareness | 2024 may- 2024 July
  General body awareness of individuals will be assessed with the Body Awareness Questionnaire (BAQ).
Neck Disability | 2024 may- 2024 July
  Neck disability index will be used to assess this parameter. The questionnaire contains 10 questions related to different activities. Each question is scored between 0 and 5. The level of disability is determined according to the total score obtained from the questionnaire. 0-4 = no disability, 5-14 = mild disability, 15-24 = moderate disability, 25- 34 = severe disability, 35 and above = total disability.
General health questionnaire | 2024 may - 2024 July
  The SF-12, which is more practical and shorter than the SF-36 but contains the same sub-dimensions as the SF-36, will be used to assess quality of life. SF-12 consists of 8 sub-dimensions and 12 items including physical functioning (2 items), physical role, body pain, general health, energy, social functioning, emotional role and mental health. The questionnaire scoring is calculated under the headings of physical and mental health, which are the two main components of general health.
weight transfer awareness | 2024 may- 2024 July
  Two scales were used to assess weight transfer awareness. Results will be recorded in kg.
neck awareness | 2024 may- 2024 July
  Individuals' neck awareness will be assessed with the Fremantle Neck Awareness Questionnaire (FreBFA).
mindfulness | 2024 may- 2024 July
  Short Form of the Five Facet Mindfulness Questionnaire (FFMQ - Short Form) will be used to assess people's mindfulness
interoception | 2024 may- 2024 July
  For the sense of interoception, the Multidimensional Assessment of Interoceptive Awareness Scale, which assesses interoceptive body awareness, will be used.
proprioception | 2024 may- 2024 July
  The Cervical Range of Motion (CROM) device is used to assess proprioception. The device assesses proprioception in 6 different directions of the neck.
verticality | 2024 may- 2024 July
  The bucket test will be used to assess subjective visual verticality, which is one of the sub-dimensions of verticality perception.
extroception | 2024 may- 2024 July
  The sense of extroception will be evaluated with the right-left hand confusion test.

SECONDARY OUTCOMES:
Pain Assessment | 2024 may- 2024 July
  Pain intensity will be assessed by Visual Analog Scale (VAS).0: I have no pain 10: I have unbearable pain In addition, pain duration and pain frequency will be questioned.
Pain self efficacy | 2024 may- 2024 July
  The Pain Self-Efficacy Questionnaire will be used to assess the confidence of people with chronic pain to perform certain tasks and behaviors despite their pain. Each item is rated on a 7-point Likert-type scale (0=not at all confident, 6=fully confident). The total score ranges from 0 to 60, with higher scores indicating greater self-efficacy for functioning despite pain.
Anxiety and Depression | 2024 may- 2024 July
  Beck Depression and Beck Anxiety scales will be used to assess depression and anxiety. Both questionnaires have 21 questions and are scored between 0-3. According to the total scores, 0-9 points in the Beck Depression Scale indicates normal level, 10-16 points indicates mild depression, 17-29 points indicates moderate depression and 30-63 points indicates severe depression. On the Beck Anxiety Scale, 0-17 points are classified as low anxiety, 18-24 points as moderate anxiety, and 25 and above points as high anxiety.
Range of motion | 2024 may- 2024 July
  Normal range of motion of the cervical region will be evaluated with the "Cervical Range of Motion" device. Active ranges of motion in flexion-extension, lateral flexion and rotation directions will be recorded with the subjec
Posture Assesment | 2024 may- 2024 July
  New York Posture Rating Scale will be used to evaluate posture. Posture changes that may occur in 13 different parts of the body including head, neck, shoulders, shoulders, back, waist, hip and ankle are observed. According to the results of the observation, five (5) points are given if the person has proper posture, three (3) points if the posture is moderately impaired, and one (1) point if there is a serious impairment. A high score means that the posture is good.
Weight transfer | 2024 may- 2024 July
  Symmetry of weight transfer to both lower extremities of the individuals in a standing upright position will be evaluated. It will be recorded in kg.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amiri Arimi S, Ghamkhar L, Kahlaee AH. The Relevance of Proprioception to Chronic Neck Pain: A Correlational Analysis of Flexor Muscle Size and Endurance, Clinical Neck Pain Characteristics, and Proprioception. Pain Med. 2018 Oct 1;19(10):2077-2088. doi: 10.1093/pm/pnx331. PMID 29304254
- [Background] Dere T, Alemdaroglu-Gurbuz I. Muscular endurance and its association with neck pain, disability, neck awareness, and kinesiophobia in patients with chronic neck pain. Somatosens Mot Res. 2024 Sep;41(3):134-141. doi: 10.1080/08990220.2023.2186390. Epub 2023 Mar 10. PMID 36897182
- See also: The Relevance of Proprioception to Chronic Neck Pain: A Correlational Analysis of Flexor Muscle Size and Endurance, Clinical Neck Pain Characteristics, and Proprioception — https://pubmed.ncbi.nlm.nih.gov/29304254/
- See also: Muscular endurance and its association with neck pain, disability, neck awareness, and kinesiophobia in patients with chronic neck pain — https://pubmed.ncbi.nlm.nih.gov/36897182/